CLINICAL TRIAL: NCT06437171
Title: The Use of Exhaled Nitric Oxide as a Predictive Marker of Allergic Reactions to Oral Food Challenge and Clinical Response of Omalizumab Treatment in Subjects With Multiple Food Allergies
Brief Title: FeNO as a Marker of Allergic Reactions to OFC and Response of OMA Treatment in Multiple FA
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AAADRS Clinical Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML45389
Record Dates: First submitted 2024-05-17; First posted 2024-05-31 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Food Allergy
Keywords: Food Allergy; Multiple Food Allergies; Biomarker
MeSH Terms: conditions — Food Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open Label Injection of Omalizumab (Other): Omalizumab dose and frequency based on baseline patient weight and total IgE
  Interventions: Biological: Omalizumab

INTERVENTIONS:
Biological: Omalizumab — Omalizumab dose and frequency based on baseline subject weight and total IgE

SUMMARY:
This is a Phase IV, open-label, single-center study to evaluate the change in FeNO as a marker of clinical response to OMA in participants with multiple FA.

DETAILED DESCRIPTION:
This is a Phase IV, open-label, single-center study to evaluate the change in FeNO as a marker of clinical response to OMA in participants with multiple FA. Twenty (20) participants will be enrolled over a 9-month enrollment period from an allergy and asthma medical specialty clinic. Should the participant meet all eligibility criteria, then following the Screening Period, the participant will be dosed with OMA and asked to continue to follow their food avoidance regimen.

Participants will return to the clinic every two weeks for 16-weeks, and then every 2 or 4-weeks (depending on dosing) for the remaining 36-weeks, for a total of 52-weeks. Primary endpoint analyses will occur at Week 16 and Week 52.

Description of XOLAIR treatment schedule:

Omalizumab will be dosed according to the OUtMATCH Study dosing. Patients will be monitored for acute hypersensitivity reactions for at least 61 minutes after the end of the injection. Epinephrine and parenteral diphenhydramine must be readily available for immediate use if required to treat a hypersensitivity reaction; site personnel must be able to detect and treat such reactions. Patients with severe hypersensitivity reactions (e.g., stridor, angioedema, life-threatening change in vital signs) must be withdrawn from study treatment.

All adverse events of systemic hypersensitivity reactions or anaphylactoid or anaphylaxis reactions must be reported within 24 hours to the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet the following criteria for study entry:

  * Able and willing to provide written informed consent from patient and parent or guardian and to comply with the study protocol.
  * Age 6 years of age or older at Visit 1
  * Documented history of food allergy to one or more of the following foods based on SPT performed at baseline visit:

    * peanut
    * milk
    * egg
    * tree nuts (Walnut/Pecan, Cashew/Pistachio, Almond, Hazelnut, Brazil nut)

Exclusion Criteria:

* Patients who meet any of the following criteria will be excluded from study entry:

  * Diagnosis of asthma requiring maintenance medication, including inhaled steroids, leukotriene modifiers, LABA/ICS, biologics medications (Intermittent asthma [Step 1] is allowed and defined according to the 2020 NAEPP guidelines (as 'asthma requiring only prn SABA use) and FEV1 < 80% of predicted normal.
  * Diagnosis of nasal polyps, cystic fibrosis or any respiratory condition that will skew normally occurring FeNO levels
  * FeNO (measured in ppb) is lower than a value expected for the age, height, and gender of the participant or inability to perform respiratory collection maneuver
  * Systemic steroids, leukotriene modifiers, or nasal steroids for any cause/diagnosis within 4 weeks of baseline
  * Biologic use, for any diagnosis, within five half-lives of Screening
  * Antibiotic use, systemic/oral/intramuscular, for any cause/diagnosis within 2 weeks of baseline
  * Active smoker, cigarette, cigar, vape, recreational, and/or prior 10 pack year history
  * Participant weight or IgE levels outside of the dosing table for OMA
  * Known history of anaphylaxis/hypersensitivity to OMA
  * Any medical condition that is serious or unstable that in the opinion of the PI could confound the study results and/or interfere with subject participation or adherence
  * Pregnant or breastfeeding, or intending to become pregnant during the study or within 60 days after the last dose of OMA
* Women of childbearing potential must have a negative serum pregnancy test result during the screening period

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
FeNO change from baseline to week 52 | 1 year
  biomarker

SECONDARY OUTCOMES:
Time to change from baseline FeNO during OFC | at baseline and at week 16
  biomarker

CONTACTS AND LOCATIONS:
Locations (1):
- AAADRS Clinical Research Center, Coral Gables, Florida, United States